CLINICAL TRIAL: NCT06346106
Title: The Diagnostic Experience of Male Rett Syndrome
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital Colorado (Other)
Collaborators: University of Colorado, Denver (Other); Vanderbilt University School of Medicine (Other); University of Alabama at Birmingham (Other); University of Pennsylvania (Other); International Rett Syndrome Foundation (Other); Rocky Mountain Rett Association (Unknown)
Responsible Party: Principal Investigator, Tim Benke, MD, Professor, Children's Hospital Colorado
Other Study IDs: 23-0075
Record Dates: First submitted 2024-02-07; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Rett Syndrome; RTT
MeSH Terms: conditions — Rett Syndrome

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: Male Rett — This study does not have an intervention. Participants of this study must be parents or caregivers to boys with Rett syndrome.

SUMMARY:
The Diagnostic Experience of Male Rett Syndrome collects information on the lived experiences of parents or caregivers to boys with Rett Syndrome. Key information examined includes the process of getting a male Rett syndrome diagnosis, your son's systems of care, and your priorities for his health needs.

Enrolled participants will complete an online survey with questions about having a son with Rett Syndrome. The Diagnostic Experience of Male Rett Syndrome study is available to parents or caregivers to boys (alive or passed) with Rett Syndrome. Compensation is not provided.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking parents (over the age of 18) of male children (all ages, alive or deceased) with confirmed genetic diagnosis of male RTT

Exclusion Criteria:

* parents of male MECP2 duplication syndrome

Ages: 0 Years to 100 Years | Sex: Male
Age Groups: Child, Adult, Older Adult
Study Population: Parents/caregivers to boys with Rett syndrome
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-05-24 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic experiences | retrospective from birth
  Qualitative interview
Attainment of developmental milestones and any regressions | retrospective from birth
  Remote survey of developmental milestones, reported in months
QI-disability | retrospective over prior month
  "QI-Disability" is a published remote survey of symptom ratings that are combined into an aggregate score of quality of life
Parent priorities for care and counseling | retrospective from birth
  Remote survey the asks parents to prioritize with a rating scale their priorities for patient care
Parenting experience | retrospective from birth
  Remote survey the asks parents to rate with a rating scale their parenting experience
Information regarding child's death, if applicable | retrospective from birth
  Questionnaire that asks parents about the details of their child's death, if applicable

SECONDARY OUTCOMES:
Family demographics | retrospective, over last 12 months
  Questionnaire
Systems of supports | retrospective, over last 12 months
  Questionnaire
Healthcare preferences | retrospective, over last 12 months
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Benke, MD, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided